CLINICAL TRIAL: NCT03614923
Title: A Phase 2, Double-Blind, Placebo-Controlled, Parallel Group, Multiple Dose Study to Investigate Etokimab (ANB020) in Adult Subjects With Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: Etokimab in Adults With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANB020-006
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-08

CONDITIONS: Chronic Rhinosinusitis
Keywords: ANB020; Etokimab; CRSwNP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Etokimab 300 mg + 150 mg Q4W (Experimental): Participants received a 300 mg loading dose of etokimab administered by subcutaneous injection at Week 0 then 150 mg etokimab by subcutaneous injection every 4 weeks (Q4W) up to Week 12 (Weeks 4, 8, and 12). Participants also used mometasone furoate nasal spray (MFNS) of 2 actuations (50 μg/actuation) in each nostril twice daily (BID).
  Interventions: Biological: Etokimab; Drug: Mometasone Furoate Nasal Spray
- Etokimab 300 mg + 150 mg Q8W (Experimental): Participants received a 300 mg loading dose of etokimab administered by subcutaneous injection at Week 0 then etokimab 150 mg by subcutaneous injection every 8 weeks (Q8W) up to Week 12 and placebo at Weeks 4 and 12. Participants also used MFNS of 2 actuations (50 μg/actuation) in each nostril BID.
  Interventions: Biological: Etokimab; Biological: Placebo; Drug: Mometasone Furoate Nasal Spray
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks up to Week 12. Participants also used MFNS of 2 actuations (50 μg/actuation) in each nostril BID.
  Interventions: Biological: Placebo; Drug: Mometasone Furoate Nasal Spray

INTERVENTIONS:
Biological: Etokimab — Administered by subcutaneous injection
  Other Names: ANB020
  Arms: Etokimab 300 mg + 150 mg Q4W; Etokimab 300 mg + 150 mg Q8W
Biological: Placebo — Administered by subcutaneous injection
  Arms: Etokimab 300 mg + 150 mg Q8W; Placebo
Drug: Mometasone Furoate Nasal Spray — Mometasone Furoate Nasal Spray (MFNS) was used from 4 weeks prior to Day 1 (Run-in period) through the end of the study. Participants used 2 actuations (50 μg/actuation) in each nostril BID, total daily dose of 400 μg. Participants intolerant to BID intranasal corticosteroids (INCS) could use the lower dose regimen of 1 actuation in each nostril BID, total daily dose of 200 μg.

SUMMARY:
A study to evaluate the safety and efficacy of multiple doses of etokimab in adults with chronic rhinosinusitis with nasal polyps.

DETAILED DESCRIPTION:
This study is a randomized, placebo controlled, double-blind, multi-dose study to assess the efficacy of two different dose regimens of etokimab compared to placebo in adults with moderate-to-severe chronic sinusitis with nasal polyposis (CRSwNP).

During the screening period, all subjects will undergo evaluation for eligibility. A centralized reader will be used to confirm the diagnosis of CRSwNP as assessed by nasal endoscopy, computed tomography (CT) scan of sinuses, and symptom scoring to reduce the risk of interpretation variation.

Participants will also be provided mometasone furoate nasal spray (MFNS) for use during the trial and are required to undergo a minimum run-in period of 20 days prior to Day 1 with approximately 80% compliance.

Participants will be randomly assigned on Day 1 to one of the three treatment arms in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of CRSwNP
* Nasal polyp score (NPS) ≥ 4 out of a maximum score for both nostrils (with at least a score of 1 for each nostril).
* 22 Item Sino-Nasal Outcome Test (SNOT-22) score > 15.
* Presence of at least two of the following symptoms prior to screening: nasal blockade/obstruction/congestion or nasal discharge (anterior/posterior nasal drip); facial pain/pressure; reduction or loss of smell
* Body mass index (BMI) of 18 to 42 kg/m^2 (inclusive) and total body weight > 50 kg (110 lb). BMI=weight (kg)/(height [m^2]).

Exclusion Criteria:

* Use of investigational drugs or prohibited therapy for this study within 8 weeks before screening or 5 half-lives, whichever is longer.
* Have experienced severe life threatening anaphylactic reactions.
* Participation in any interventional study for the treatment of CRSwNP in the 3 months before screening.
* If female, is pregnant or lactating, or intend to become pregnant during the study period.
* History (or suspected history) of alcohol or substance abuse.
* Current smokers or former smokers with a smoking history of ≥ 10 pack years. If a patient has less than 10 pack years smoking history, he or she should have quit smoking at least 2 months before screening to enroll in the study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SM_ANB020-006@syneoshealth.com, Study Director — AnaptysBio, Inc.
Locations (28):
- United States (28):
  - Asthma & Allergy Institute, Little Rock, Arkansas
  - Alliance Research Institute, Canoga Park, California
  - DaVinci Research, Roseville, California
  - Sacramento Ear Nose and Throat Surgical and Medical Group Inc. - SacENT, Sacramento, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - Colorado Allergy Asthma Centers, Denver, Colorado
  - Intermed Medical Research Center, Miami, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Clinical Research Consultants of Atlanta, Suwanee, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Chicago ENT, Chicago, Illinois
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Chesapeake Clinical Research Inc., Baltimore, Maryland
  - ENT and Allergy Associates ENTA LLP, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, Matthews, North Carolina
  - Ohio Sinus Institute, Dublin, Ohio
  - Allergy Asthma Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy Asthma and Immunology Center P.C., Tulsa, Oklahoma
  - Central States Research, LLC, Tulsa, Oklahoma
  - National Allergy and Asthma Research, North Charleston, South Carolina
  - Fort Worth ENT Berkson Medical, Fort Worth, Texas
  - Ear Nose and Throat Associates of Texas, McKinney, Texas
  - Intermountain Ear Nose Throat Specialist, Draper, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Eastern Virginia Medical School EVMS Medical Group, Norfolk, Virginia
  - Bellingham Asthma Allergy Immunology Clinic, Bellingham, Washington
  - Allergy, Asthma Sinus Center, SC, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 sites in the United States.
Pre-assignment Details: All participants entered a run-in period of between 20 and 31 days on mometasone furoate nasal spray (MFNS) of two actuations (50 μg/actuation) in each nostril twice daily (BID) prior to Day 1.
  Eligible participants were randomly assigned on Day 1 to one of three treatment arms in a 1:1:1 ratio. Randomization was stratified by asthma comorbidity.
Period: Overall Study
Arm/Group | Etokimab 300 mg + 150 mg Q4W | Etokimab 300 mg + 150 mg Q8W | Placebo
Started | 35 | 35 | 35
Completed | 30 | 30 | 30
Not Completed | 5 | 5 | 5
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Non-compliance | 0 | 1 | 0
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Etokimab 300 mg + 150 mg Q4W: Participants received a 300 mg loading dose of etokimab administered by subcutaneous injection at Week 0 then 150 mg etokimab by subcutaneous injection Q4W up to Week 12 (Weeks 4, 8, and 12). Participants also used MFNS of 2 actuations (50 μg/actuation) in each nostril BID.
- Etokimab 300 mg + 150 mg Q8W: Participants received a 300 mg loading dose of etokimab administered by subcutaneous injection at Week 0 then etokimab 150 mg by subcutaneous injection Q8W up to Week 12 and placebo at Weeks 4 and 12. Participants also used MFNS of 2 actuations (50 μg/actuation) in each nostril BID.
- Total: Total of all reporting groups
Arm/Group | Etokimab 300 mg + 150 mg Q4W | Etokimab 300 mg + 150 mg Q8W | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (14.82) | 48.2 (10.28) | 49.5 (12.68) | 49.0 (12.62)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 32 | 35 | 31 | 98
  >=65 years | 3 | 0 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 9 | 29
  Male | 27 | 23 | 26 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 5 | 13
  Not Hispanic or Latino | 29 | 33 | 30 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 5 | 12
  White | 33 | 29 | 30 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Nasal Polyp Score (NPS) [Mean (Standard Deviation); unit: score on a scale] — Nasal endoscopies were performed using centralized imaging data assessments and scored by an independent reviewer. Nasal polyps were scored from 0 (no polyps) to 4 (polyps causing complete obstruction of the inferior nasal cavity).
  The bilateral NPS score is the sum of the right and left nostril scores, hence the total NPS ranges from 0 to 8 (worst). Population: The full analysis set included all randomized participants who received at least one dose of etokimab or placebo, and had a Baseline and at least one post-Baseline NPS and/or SNOT-22 score up to Week 16.
  score on a scale
    number analyzed (Participants) | 34 | 35 | 35 | 104
    (all) | 5.4 (1.58) | 5.2 (2.01) | 5.7 (1.86) | 5.4 (1.83)
Sino-Nasal Outcome Test (SNOT-22) Score [Mean (Standard Deviation); unit: score on a scale] — SNOT-22 is a 22-item outcome measure on a 5-category scale that assesses symptoms and social/emotional consequences of rhinosinusitis. Each item is scored from 0 (No problem at all) to 5 (Problem as bad as it can be), and the total score ranges from 0 to 110. Higher SNOT-22 scores are indicative of greater impact of rhinosinusitis on quality of life. Population: The full analysis set included all randomized participants who received at least one dose of etokimab or placebo, and had a Baseline and at least one post-Baseline NPS and/or SNOT-22 score up to Week 16.
  score on a scale
    number analyzed (Participants) | 34 | 35 | 35 | 104
    (all) | 51.4 (19.73) | 53.9 (23.67) | 56.9 (21.69) | 54.1 (21.78)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Nasal Polyp Score (NPS) to Week 16
Description: Nasal polyps were evaluated by nasal endoscopy using centralized imaging data assessments scored by an independent reviewer.
  Each nostril was scored on a scale from 0 to 4, where a score of 0 means no polyps, and a score of 4 means the presence of polyps causing complete obstruction of the inferior nasal cavity.
  The bilateral NPS score is the sum of the right and left nostril scores, and hence the total NPS value is between 0 and 8 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Etokimab 300 mg + 150 mg Q4W | Etokimab 300 mg + 150 mg Q8W | Placebo
Number analyzed (Participants) | 29 | 33 | 31
score on a scale | -0.87 (0.225) | -0.89 (0.221) | -0.49 (0.225)
Statistical Analysis 1: Comparison: Etokimab 300 mg + 150 mg Q4W vs Placebo; A general linear mixed effects model with repeated measures (MMRM) was used including the change from Baseline in NPS as dependent variable; treatment group, stratification factor, time (Weeks 4, 8, 12, and 16), treatment by stratification factor, and treatment by time interaction as fixed effect factors; Baseline NPS as covariate; and subject as random effect; Test type: Superiority — Statistical significance for the co-primary efficacy endpoints would be declared if both p-values for the tests of the individual hypotheses were < 0.05; p = 0.2364, General linear MMRM — Testing was conducted in a hierarchical manner such that the comparison of etokimab Q4W versus placebo was conducted first. If the results of this comparison were statistically significant, the etokimab Q8W treatment arm would be compared to placebo; Least Squares (LS) Mean Difference = -0.38, 95% CI 2-sided [-1.01 to 0.25], Standard Error of Mean 0.319
Statistical Analysis 2: Comparison: Etokimab 300 mg + 150 mg Q8W vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Statistical significance for the co-primary efficacy endpoints was to be declared if both p-values for the tests of the individual hypotheses were < 0.05; p = 0.2024, General linear MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.41, 95% CI 2-sided [-1.03 to 0.22], Standard Error of Mean 0.316

2. Primary Outcome: Change From Baseline in Sino-Nasal Outcome Test-22 (SNOT-22) Score at Week 16
Description: SNOT-22 is a 22-item outcome measure on a 5-category scale that assesses symptoms and social/emotional consequences of rhinosinusitis. Each item is scored from 0 (No problem at all) to 5 (Problem as bad as it can be), and the total score ranges from 0 to 110. Higher SNOT-22 scores are indicative of greater impact of rhinosinusitis on quality of life. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set participants with available data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Etokimab 300 mg + 150 mg Q4W | Etokimab 300 mg + 150 mg Q8W | Placebo
Number analyzed (Participants) | 30 | 33 | 31
score on a scale | -22.97 (3.084) | -18.34 (3.077) | -16.32 (3.112)
Statistical Analysis 1: Comparison: Etokimab 300 mg + 150 mg Q4W vs Placebo; A general linear mixed effects model with repeated measures (MMRM) was used including the change from Baseline in SNOT-22 as dependent variable; treatment group, stratification factor, time (Weeks 4, 8, 12, and 16), treatment by stratification factor, and treatment by time interaction as fixed effect factors; Baseline SNOT-22 as covariate; and subject as random effect; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.1330, General linear MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -6.64, 95% CI 2-sided [-15.34 to 2.06], Standard Error of Mean 4.383
Statistical Analysis 2: Comparison: Etokimab 300 mg + 150 mg Q8W vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.6464, General linear MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -2.01, 95% CI 2-sided [-10.70 to 6.67], Standard Error of Mean 4.375

3. Secondary Outcome: Change From Baseline in Eosinophil Count
Time Frame: Baseline, Week 16, and Week 24
Population: Safety analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Etokimab 300 mg + 150 mg Q4W | Etokimab 300 mg + 150 mg Q8W | Placebo
Number analyzed (Participants) | 35 | 35 | 35
10^9 cells/L
  Baseline | 0.437 (0.2546) | 0.350 (0.2038) | 0.434 (0.2490)
  Change from Baseline at Week 16: number analyzed (Participants) | 30 | 33 | 30
  Change from Baseline at Week 16 | -0.162 (0.1717) | -0.117 (0.1718) | -0.020 (0.1843)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 3 | 28
  Change from Baseline at Week 24 | -0.038 (0.2451) | -0.029 (0.1674) | 0.019 (0.2151)

ADVERSE EVENTS:
Time Frame: From first dose of study medication on Day 1 until Week 16, or up to 28 days after the last dose of study medication for participants who discontinued treatment earlier than Week 16.
Arm/Group | Etokimab 300 mg + 150 mg Q4W | Etokimab 300 mg + 150 mg Q8W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 8/35 | 8/35 | 6/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etokimab 300 mg + 150 mg Q4W (N=35) | Etokimab 300 mg + 150 mg Q8W (N=35) | Placebo (N=35)
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etokimab 300 mg + 150 mg Q4W (N=35) | Etokimab 300 mg + 150 mg Q8W (N=35) | Placebo (N=35)
Sinusitis (Infections and infestations) | 2 | 5 | 4
Headache (Nervous system disorders) | 1 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Injection site erythema (General disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is 18 months since study completion. Then, Investigator can publish if manuscript is submitted to Sponsor 90 days prior to submission. Sponsor may require the Investigator to remove specifically identified Confidential Information (other than Trial Data) and/or to delay the proposed publication for an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (2):
  • Study Protocol (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03614923/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03614923/SAP_001.pdf